CLINICAL TRIAL: NCT05404724
Title: Study on the Pharmacokinetic Effects of Single-centered, Open, Single-arm, Fixed-sequence Itraconazole on SHR0302 Tablets in Healthy Subjects
Brief Title: Study on the Pharmacokinetic Effect of Itraconazole on SHR0302 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR0302-110
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: itraconazole and SHR0302 tablets are used in combination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): itraconazole and SHR0302 tablets
  Interventions: Drug: itraconazole、 SHR0302 tablets

INTERVENTIONS:
Drug: itraconazole、 SHR0302 tablets — Itraconazole 7 times and SHR0302 tablets twice. On the 8th day of this, itraconazole and SHR0302 tablets were taken simultaneously.

SUMMARY:
To evaluate the effect of oral itraconazole on the pharmacokinetics of SHR0302 in healthy subjects.

To evaluate the safety and tolerability of oral SHR0302 and itraconazole monotherapy and combination use in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form prior to the commencement of activities related to this trial, be able to understand the procedures and methods of this trial, and be willing to strictly comply with the clinical trial protocol to complete this trial;
2. Age 18 to 45 years (inclusive, subject to the signing of informed consent), healthy male;
3. Body mass ≥ 50 kg and body mass index (BMI): 19 to 26 kg/m2 (both ends included);
4. Be able to communicate well with the investigators and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Those who have participated in clinical trials of any drug and medical device within three months before the first administration or who are still in the follow-up period of a clinical study or 5 half-life periods of the test drug before screening (whichever is longer), the participant in the clinical trial is defined as: those who have signed informed consent for clinical trials and have used the test drugs (including placebo) or experimental medical devices;
2. Those who have chronic or active gastrointestinal diseases such as esophageal diseases, gastritis, gastric ulcers, enteritis, active gastrointestinal bleeding or gastrointestinal surgery within three years and the researchers believe that there is still clinical significance;
3. Those who have a history of respiratory system, cardiovascular system, endocrine system, urinary system, nervous system, hematology, immunology (including personal or family history of hereditary immunodeficiency), metabolic abnormalities, etc., and the researcher believes that there is still clinical significance;
4. Patients with a history of ventricular dysfunction;
5. Have any history of systemic inflammatory diseases, autoimmune diseases, recurrent herpes zoster, disseminated herpes zoster, and disseminated herpes simplex;
6. Those who have a history of tuberculosis (TB) within half a year before the first administration;
7. Infections or other acute diseases that need to be treated with antimicrobials (viral, bacterial, fungal, parasitic infections) within 4 weeks before the first administration of the drug are judged by the researchers to be unsuitable for participating in the trial;
8. Allergic to the study drug (SHR0302 tablets and itraconazole capsules) or any ingredient in the study drug, or have a history of allergy to drugs, food or other substances;
9. Those who cannot tolerate intravenous puncture or have a history of blood sickness and needle sickness;
10. Those who have undergone surgery that the researchers judge will affect the absorption, distribution, metabolism and excretion of the drug within 6 months before the first administration; or have undergone surgery within 4 weeks before the first administration; or those who plan to perform surgical operations during the trial period;
11. Those who have used any drugs (including Chinese herbal medicines, health care products, etc.) within 14 days before the first administration, or those who plan to take drugs or health care products that are not experimental in this study during the trial period;
12. Any drug or food that has been used within 30 days prior to the first administration is an inhibitor or inducer of the cytochrome P4503A4 enzyme (CYP3A4), as detailed in Annex 2;
13. those who have received BCG vaccine within 12 months prior to the first dose, or who have been vaccinated or exposed to other live vaccines or live attenuated vaccines within 3 months prior to the first dose, or who plan to be vaccinated during the trial;
14. those who donate blood or lose a large amount of blood (> 400 mL) within 3 months before the first administration, those who receive blood transfusions or use blood products, or those who intend to donate blood or blood components during the trial period or within 3 months after the end of the test;
15. Drug abusers or those who have used soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the first administration of drugs;
16. Smokers or smokers with more than 5 cigarettes per day in the 3 months before the first administration, or who cannot stop using any tobacco-based products during the trial;
17. Alcoholics or regular drinkers in the 6 months prior to the first administration of the drug, i.e. those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits or 150 mL of wine with an alcohol content of 45 mL); or are unwilling to stop drinking alcohol or any alcoholic products during the trial;
18. those who drink excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day, or those who do not agree to stop drinking tea, coffee and/or caffeinated beverages during the trial period;
19. those who have eaten any beverage or food containing grapefruit within 7 days before the first administration, or any beverage or food containing methylxanthine, such as coffee, tea, cola, chocolate, etc., within 48 hours before the first administration; or do not agree to stop eating the above diet during the trial period;
20. Those who have special requirements for diet and cannot comply with the unified diet;
21. During the test period, strenuous exercise cannot be stopped, or there are other factors that may affect the absorption, distribution, metabolism, excretion and other factors of the drug;
22. Volunteers who have a fertility plan, a sperm donation and egg donation plan during the trial period and 6 months after the end of the trial, or are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, contraceptive rings, partner sterilization, etc.);
23. Abnormal clinical significance of physical examination, electrocardiogram, vital signs, color ultrasound of the heart and abdomen, chest orthostatic film, and laboratory examination (subject to the judgment of the clinician);
24. ECG examination QTc>440 ms;
25. Glomerular filtration rate (eGFR）<90 mL/min/1.73m2(Adopt simplified renal disease dietary adjustments (MDRDformula calculation,eGFR=186×[serum creatinine value (mg/dL）]-1.154×[Age (years)]-0.203oreGFR=186×[serum creatinine value (μmol/L）×0.01131]-1.154×[Age (years)]-0.203）;
26. Positive uremic screen test;
27. Positive alcohol breath test;
28. Volunteers may not be able to complete this study for other reasons or have other reasons that the researchers judge that they are not suitable to participate in the trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
SHR0302 and its main metabolite AUC0-t | day 1 to day 11
SHR0302 and its main metabolite AUC0-inf | day 1 to day 11
SHR0302 and its main metabolite Cmax | day 1 to day 11

SECONDARY OUTCOMES:
SHR0302 and its main metabolite Tmax (SHR0302 only) | day 1 to day 11
SHR0302 and its main metabolite t1/2 (SHR0302 only) | day 1 to day 11
SHR0302 and its main metabolite CL/F (SHR0302 only) | day 1 to day 11
SHR0302 and its main metabolite Vz/F (SHR0302 only) | day 1 to day 11
Adverse events | Day 1 to Day 17

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided